CLINICAL TRIAL: NCT05830240
Title: A Clinical Safety and Efficacy Study on Oncolytic Virus Injection (R130) for the Treatment of Relapsed/Refractory Head and Neck Cancer
Brief Title: A Clinical Study on Oncolytic Virus Injection (R130 OV) for the Treatment of Relapsed/Refractory Head and Neck Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Yunying Medical Technology (Industry)
Collaborators: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHWG-R130-HNC
Record Dates: First submitted 2023-03-31; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Cancer; Esophageal Cancer; Otorhinolaryngologic Neoplasms; Ear Cancer; Nose Cancer; Laryngeal Cancer; Pharyngeal Cancer
Keywords: Oncolytic virus; Herpes simplex virus type 1
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms; Otorhinolaryngologic Neoplasms; Ear Neoplasms; Nose Neoplasms; Laryngeal Neoplasms; Pharyngeal Neoplasms | interventions — Oncolytic Virotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R130 Treatment Group (Experimental): Every 7-14 days,1-2 ml R130 （concentration of 1x10^8 plaque-forming Units/mL,PFU/mL）will be injected intratumoral in patients with relapsed/refractory head and neck cancer
  Interventions: Drug: Recombinant oncolytic herpes simplex virus type 1 (R130)

INTERVENTIONS:
Drug: Recombinant oncolytic herpes simplex virus type 1 (R130) — R130, a modified herpes simplex virus-Ⅰ (HSV-1) containing the gene coding for anti-CD3 scFv/CD86/PD1/HSV2-US11
  Other Names: Oncolytic virus

SUMMARY:
9 participants are expected to be enrolled for this open，single-armed clinical trial to evaluate the safety and efficacy of the recombinant herpes simplex virus Ⅰ, R130 in patients with relapsed/refractory head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with head and neck cancer clearly diagnosed by histology and/or cytology, without systematic metastasis, and failure of standard treatment.
2. Age 18 to 75 years.
3. No absolute or relative centasis contraindiction，have at least one measurable lesion (according to RECIST 1.1 criteria) that is amenable to intratumoral drug delivery.
4. No severe functinonal falure of heart, brain, liver, kidney and lung.
5. Subjects with ECOG score of 0-2, and expected survival of 3 months or more.
6. No evidence of clinically significant immunosuppression.
7. Patients must have the following hematologic parameters, Coagulation functions and hepatic and renal function during the screening period:

   * White Blood Cell (WBC)≥3.0×10^9/L；
   * Absolute Lymphocyte Count (ANC)≥1.5×10^9/L;
   * Platelet≥100×10^9/L；
   * Prothrombin time (PT) or activated Partial Thromboplastin Time（APTT）≤1.5×ULN;
   * Serum Creatinine (Scr)≤1.5×ULN
   * Alanine aminotransferase(AST/ALT) ≤3×ULN;
   * Total Bilirubin(TBIL)≤1.5×ULN.
8. Be able to understand and sign the informed consent document;
9. Be able to stick to follow-up visit plan and other requirements in the agreement.

Exclusion Criteria.

1. With a history of allergy to similar drugs.
2. With hematological diseases, malignant tumors of the central nervous system, or combined with other malignant tumors.
3. pregnancy, breast feeding.
4. Current active hepatitis B, active hepatitis C, immunodeficiency virus or other active infection of clinical significance.
5. Impaired function of important organs or a history of organ transplantation.
6. Receiving antiherpes simplex virus therapy such as acyclovir, ganciclovir, vancomycin, and acepromazine within 4 weeks.
7. Have had antitumor therapy, including endocrine, chemotherapy, radiotherapy, targeted therapy, immunotherapy and antitumor herbal therapy,4 weeks prior to the first dose.
8. Have had any serious adverse reactions associated with immunotherapy and have not recovered to CTCAE 5.0 grade rating 0 or 1 level of toxicity after previous antineoplastic therapy.
9. Subjects with any severe and/or uncontrolled disease, including: a) poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); b) suffering from class I or higher myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥ 470 ms and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification); c) active or uncontrolled severe infection (≥ CTCAE grade 2 infection); d) Patients with previous organ transplantation, bone marrow transplantation (hematopoietic stem cell transplantation) and severe immune deficiency; e) Urine routine suggesting urine protein ≥++ and confirmed 24-hour urine protein quantification > 1.0 g.
10. Patients with past history of type I diabetes mellitus.
11. Severe abnormalities in thyroid and cortisol testing; active, known or suspected autoimmune disease requiring systemic therapy.
12. Patients with active bleeding or severe coagulation dysfunction.
13. Researchers considering the test subject as having a history of other severe systemic diseases, or other reasons inappropriate for the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Safety Profile Measured by Grade ≥3 CTCAE v5.0 | Up to 6 months
  To characterize the safety profile of R130 injection in patients with relapsed/refractory head and neck cancer as measured by the incidence of Grade ≥ 3 Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0)
Systemic immune response | Up to 6 months
  Detection of increased systemic immune Response markers in sera (IL2,IL4,IL6,IL8,IL10,TNFa，IFNγ, etc.) and peripheral blood mononuclear cells by multi-Color fluorescence-activated cell sorting (FACS)

SECONDARY OUTCOMES:
Disease Assessment for Disease Control Rate | Every 10 weeks for 12 months
  Evaluate the efficacy endpoints of DCR by the investigator with RECIST v1.1 and iRECIST
Disease Assessment for Duration of Response | Every 10 weeks for 12 months
  Evaluate the efficacy endpoints of DOR by the investigator with RECIST v1.1 and iRECIST
Quality of Life Assessment | Every 6 weeks for 12 months
  Evaluate with EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wu, Phd, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No